CLINICAL TRIAL: NCT00395486
Title: A 6-week, Randomised, Open-label, Parallel Group, Multi-centre Study to Compare the Efficacy of Rosuvastatin 10mg With Atorvastatin 10mg in the Treatment of Metabolic Syndrome Subjects With Raised LDL-C
Brief Title: ROMEO (Rosuvastatin in Metabolic syndrOme)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D3560L00061; ROMEO
Record Dates: First submitted 2006-11-01; First posted 2006-11-03 (Estimated); Results first posted 2011-06-16 (Estimated); Last update posted 2011-07-11 (Estimated); Status verified 2011-06

CONDITIONS: Metabolic Syndrome X
Keywords: rosuvastatin; lipoprotein; metabolic syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Rosuvastatin Calcium; Atorvastatin

ARMS (2):
- Rosuvastatin (Experimental)
  Interventions: Drug: Rosuvastatin
- Atorvastatin (Active Comparator)
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Rosuvastatin — 10mg
  Other Names: Crestor
  Arms: Rosuvastatin
Drug: Atorvastatin — 10mg
  Arms: Atorvastatin

SUMMARY:
The primary objective of this study is to compare the effect of rosuvastatin 10mg with atorvastatin 10mg after 6 weeks of treatment in the ratio of ApoB/ApoA1 in subjects with metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Presence of 3 or more of the following criteria;

  * Abdominal obesity (men >90cm women >80cm)
  * Triglycerides ≥ 150 mg/dL
  * HDL-C: men < 40 mg/dL, women < 50 mg/dL
  * BP ≥130/≥85 mmHg or anti-hypertensive treatment
  * Fasting blood glucose ≥100 mg dL or anti-diabetic treatment
* Elevated LDL-C ;

  * ≥130 mg/dL to < 220 mg/dL in lipid lowering agent naive subjects
  * ≥100 mg/dL to < 200 mg/dL in subjects who have taken a lipid lowering drug(s) within 4 weeks of visit 1.
* Triglyceride < 500 mg/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2006-09; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: JoonWoo Bahn, MD, Study Director — AstraZeneca
Locations (3):
- South Korea (3):
  - Research Site, Pusan
  - Research Site, Seoul
  - Research Site, Suwon

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 613 subjects were enrolled in the study at 13 centres, of whom 258 were randomized to treatment with rosuvastatin (n=132) or atorvastatin (n=126). Subjects were recruited throughout South Korea from September 2006 to June 2008.
Pre-assignment Details: Enrolled patients to be randomized should complete 6-week dietary run-in periods. Also, LDL level should be ≥ 130mg/dl & < 220mg/dl and triglyceride should be < 500mg/dl.
Period: Overall Study
Arm/Group | Rosuvastatin | Atorvastatin
Started | 132 (Randomized subjects) | 126 (Randomized subjects)
Completed | 126 (Completed subjects) | 121 (Completed subjects)
Not Completed | 6 | 5
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 5 | 2
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rosuvastatin | Atorvastatin | Total
Number analyzed (Participants) | 132 | 126 | 258
Age Continuous [Mean (Standard Deviation); unit: years]
  18 years | 57.5 (10.0) | 60.4 (9.0) | 58.9 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 88 | 162
  Male | 58 | 38 | 96

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in Ratio of Apolipoprotein (ApoB/ApoA1) at Week 6
Description: Samples for evaluation from all investigational sites will be delivered by courier to the central laboratory within 24 hours of blood being drawn. This outcome will be calculated by using the result of ApoB and ApoA1.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Rosuvastatin | Atorvastatin
Number analyzed (Participants) | 127 | 122
percent change | -44.40 (14.70) | -36.50 (14.10)

2. Secondary Outcome: Percentage of Subjects Reaching Their LDL-C Target Goal
Description: Based on NCEP ATP III guideline, calculate the percentage of subjects reaching their LDL-C target goal. LDL-C target goals are <70mg/dl, <100mg/dl and <130mg/dl according to their baseline conditions (presence of Coronary heart disease and risk factors and grade of Framingham 10-Year risk).
Time Frame: Baseline and 6 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Rosuvastatin | Atorvastatin
Number analyzed (Participants) | 127 | 122
percentage of participants | 88.20 | 75.40

3. Secondary Outcome: Percentage of Subjects Reaching Their Low-Density Lipoprotein-C (LDL-C) and Non High-Density Lipoprotein-C (HDL-C) Target Goal
Description: Based on NCEP ATP III guideline, calculate the percentage of subjects reaching their LDL-C & non HDL-C target goal.
Time Frame: Baseline and 6 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Rosuvastatin | Atorvastatin
Number analyzed (Participants) | 52 | 48
percentage of participants | 78.80 | 66.70

4. Secondary Outcome: Percentage Change of Glucose Level
Description: Using laboratory test, mean change of glucose level was investigated.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Rosuvastatin | Atorvastatin
Number analyzed (Participants) | 127 | 122
Percentage change | -0.60 (10.10) | 2.78 (13.90)

5. Secondary Outcome: Percentage Change of Insulin Resistance Using HOMA-R
Description: HOMA-R was calculated using insulin and glucose levels derived by laboratory test. The formula is as following: HOMA-R = insulin* glucose/22.5
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Rosuvastatin | Atorvastatin
Number analyzed (Participants) | 127 | 122
percentage change | 28.00 (95.20) | 50.30 (287.50)

6. Secondary Outcome: Percentage Change of Insulin Resistance Using QUICKI
Description: QUICKI was calculated using insulin and glucose levels derived by laboratory test. The formula is as following: QUICKI = 1/[log(insulin) + log(glucose)].
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Rosuvastatin | Atorvastatin
Number analyzed (Participants) | 127 | 122
percentage change | -1.27 (13.90) | -1.03 (15.00)

7. Secondary Outcome: Percentage Reduction of Low-Density Lipoprotein-C (LDL-C)
Description: Calculate the percentage reduction of LDL-C
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: percentage reduction
Arm/Group | Rosuvastatin | Atorvastatin
Number analyzed (Participants) | 127 | 122
percentage reduction | -45.50 (15.10) | -37.90 (13.40)

8. Secondary Outcome: Percentage Change of Total Cholesterol (TC)
Description: Calculate the percentage change of total cholesterol level
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Rosuvastatin | Atorvastatin
Number analyzed (Participants) | 127 | 122
percentage change | -34.10 (11.20) | -28.80 (10.90)

9. Secondary Outcome: Percentage Change of High-Density Lipoprotein-C (HDL-C)
Description: Calculate the percentage change of HDL-C level
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Rosuvastatin | Atorvastatin
Number analyzed (Participants) | 127 | 122
percentage change | 9.90 (16.40) | 8.20 (18.70)

10. Secondary Outcome: Percentage Change of Triglycerides (TG)
Description: Calculate the percentage change of Triglycerides.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Rosuvastatin | Atorvastatin
Number analyzed (Participants) | 127 | 122
percentage change | -17.20 (33.90) | -15.10 (43.50)

11. Secondary Outcome: Percentage Change of Apolipoprotein A1 (ApoA1)
Description: Calculate the percentage change of Apolipoprotein A1
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Rosuvastatin | Atorvastatin
Number analyzed (Participants) | 127 | 122
percentage change | 8.50 (12.40) | 4.20 (13.30)

12. Secondary Outcome: Percentage Change of Apolipoprotein B (ApoB)
Description: Calculate the percentage change of apolipoprotein B
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Rosuvastatin | Atorvastatin
Number analyzed (Participants) | 127 | 22
percentage change | -40.50 (14.10) | -34.60 (13.00)

ADVERSE EVENTS:
Arm/Group | Rosuvastatin | Atorvastatin
Serious Adverse Events (participants affected / at risk) | 0/129 | 4/124
Other Adverse Events (participants affected / at risk) | 0/129 | 0/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rosuvastatin (N=129) | Atorvastatin (N=124)
Arrhythmia (Cardiac disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Gastroenteritis (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less